CLINICAL TRIAL: NCT03116828
Title: Efficacy and Safety of Eslicarbazepine Acetate as First Add-on to Levetiracetam or Lamotrigine Monotherapy or as Later Adjunctive Treatment for Subjects With Uncontrolled Partial-onset Seizures: A Multicenter, Open-label, Non-randomized Trial
Brief Title: A Study of a Drug to be Used in Addition With Another Drug to Treat Adults With Uncontrolled Partial-onset Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 093-701
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Epilepsy With Partial On-set Seizures
Keywords: epilepsy; seizures; partial on-set seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — eslicarbazepine acetate

STUDY DESIGN:
Intervention Model Description: Arm 1 (ESL as first add-on) Arm 2 (ESL as later add-on)
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- eslicarbazepine acetate (arm 1) (Experimental): eslicarbazepine acetate (as first add-on)mg/day as medically indicated at the discretion of Investigator up to a maximum dose of 1200 mg/day (Canadian sites) or 1600 mg/day (US sites)
  Interventions: Drug: Eslicarbazepine acetate
- eslicarbazepine acetate (arm 2) (Experimental): eslicarbazepine acetate (as later add-on)
  Interventions: Drug: Eslicarbazepine acetate

INTERVENTIONS:
Drug: Eslicarbazepine acetate — eslicarbazepine acetate tablets, taken once daily. Subjects begin 2-week Titration Phase starting on Day 1 (Week 1), by initiating treatment with ESL 400 mg/day. Subjects titrate to minimum dose of 800 mg/day for the 24-week Maintenance Phase beginning at Week 3. In the Maintenance Phase, subjects may titrate in weekly increments of 400 mg/day as medically indicated at the discretion of Investigator up to a maximum dose of 1200 mg/day (Canadian sites) or 1600 mg/day (US sites)
  Other Names: Aptiom; ESL; SEP-0002093; BIA-2-093
Drug: Eslicarbazepine Acetate — eslicarbazepine acetate acetate tablets, taken once daily. Subjects begin 2-week Titration Phase starting on Day 1 (Week 1), by initiating treatment with ESL 400 mg/day. Subjects titrate to minimum dose of 800 mg/day for the 24-week Maintenance Phase beginning at Week 3. In the Maintenance Phase, subjects may titrate in weekly increments of 400 mg/day as medically indicated at the discretion of Investigator up to a maximum dose of 1200 mg/day (Canadian sites) or 1600 mg/day (US sites)
  Other Names: Aptiom; ESL; SEP-0002093; BIA-2-093

SUMMARY:
A study of a drug to be used in addition with another drug to treat adults with Uncontrolled Partial-onset Seizures

DETAILED DESCRIPTION:
This is a 31-week, multicenter, 2-arm, prospective, open-label, non-randomized, Phase 4 study of eslicarbazepine acetate (ESL) as adjunctive therapy in adult subjects with a diagnosis of epilepsy with POS. Two groups of ESL-naïve subjects will be evaluated. The groups are defined as follows:

* Arm 1 (ESL as first add-on): This group will include subjects who have been maintained on a regimen consisting of a stable dose of LEV or LTG for at least 1 month (28 days) prior to screening and who have not used any adjunctive treatment.
* Arm 2 (ESL as later add-on): This group will include subjects who have been maintained on a regimen consisting of a stable dose of 1-2 AEDs (excluding oxcarbazepine [OXC]) for at least 1 month (28 days) prior to screening and who have used adjunctive treatment in the past.

The Arm 1 subjects will allow an assessment of the efficacy and safety of ESL in subjects who are early in the course of their disease and being treated with one of the most common first line AEDs.

The subjects in Arm 2 are similar to the subject population in the ESL Phase 3 adjunctive epilepsy studies, treatment-resistant subjects who are later in the course of their disease. The inclusion of these subjects in the present study will provide an assessment of the efficacy and safety of ESL as a later adjunctive therapy in a real world clinical setting.

In addition, this study will provide data from both Arm 1 and Arm 2 for several behavioral, mood-related, and QOL-related assessments that were not evaluated in the ESL Phase 3 adjunctive epilepsy program.

The study will consist of a Screening Phase of 1 to 2 weeks, followed by a 2-week Titration Phase, a 24-week Maintenance Phase, and a Safety Follow-up/Taper Phase of 4 weeks. The last visit in the Maintenance Phase (Visit 9) is considered the End of Study (EOS) visit

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 18 years of age.
2. Subject is willing and able to sign informed consent.
3. Subject has a documented diagnosis of epilepsy with simple POS with a motor component or complex POS with or without secondarily generalized seizures as defined in the Classification of Seizures of the International League Against Epilepsy
4. Subject has a documented electroencephalogram within 10 years prior to screening.
5. Subject has had at least 3 POS during previous six months.
6. Subject has had a sufficient number of seizures at time of enrollment to justify adjunctive therapy, as determined by the Investigator.
7. Subjects are required to be ESL-naïve AND

   1. Maintained on a stable LEV or LTG regimen for at least 1 month (28 days) prior to screening with no history of adjunctive treatment (for Arm 1, ESL as first add-on).

      OR
   2. Maintained on a stable dose of 1-2 AEDs (excluding OXC) for at least 1 month (28 days) prior to screening and who have had prior adjunctive treatment (for Arm 2, ESL as later add-on).
8. If the subject is treated with any stimulation device for epilepsy Vagal Nerve Stimulation (VNS), Responsive Neurostimulator (RNS), or similar, the device must have been implanted at least 6 months before screening and the device parameters must be documented as stable for at least 1 month prior to screening. (Note: These devices will not be counted as concomitant AED).
9. Except for epilepsy, subject is judged to be in general good health based on medical history, physical examination findings, and clinical laboratory

Exclusion Criteria:

1. Subjects with a prior exposure to ESL.
2. Subjects currently being treated with OXC.
3. Subject with a history of allergic reaction to OXC or CBZ, or a history of serious allergic reaction (Stevens-Johnson syndrome, Drug Reaction with Eosinophilia and Systemic Symptoms or similar) to any AED, or a history of serious allergic reactions to other medications.
4. Subjects who have taken warfarin, felbamate, vigabatrin, or perampanel, (unless at stable dose with safety testing for ≥ 1 year) within a 4-week period prior to screening.
5. Subjects taking ezogabine

   .
6. Subject has taken any medication prohibited for this protocol within 4 weeks prior to Screening
7. Subjects using benzodiazepines on more than an occasional basis (defined as more than 2 times per week), except when used chronically as an AED
8. Seizure disorder characterized primarily by simple POS without motor signs.
9. Subject has a history of primarily generalized seizures (eg, myoclonic, absence, tonic).
10. Subject has a history of status epilepticus or cluster seizures (ie, 3 or more seizures within 30 minutes) within the 3 months prior to screening.
11. Subject has had seizures of psychogenic origin or purely subjective seizures within the last 2 years.
12. Subject has had seizures too close to count accurately.
13. Subject has a known progressive structural central nervous system (CNS) lesion, progressive encephalopathy or any other condition that may result in epilepsy secondary to a cerebral abnormality.
14. Subject whose current seizures are related to an acute medical illness or other non-epileptic origin.
15. Subjects of Asian ancestry will be excluded if they are carriers of HLA-B*1502. Either:

    1. Subject must give written informed consent for genotyping, and test negative. OR
    2. Subjects must provide documentation of prior testing confirming non-carrier status.
16. Subject has a major medical illness other than epilepsy that would prevent safe participation in this study, at the discretion of the Investigator, including (but not limited to) cardiac disease, thyroid disease, hepatic or renal impairment, endocrine or metabolic disease, gastrointestinal disease, or hematologic disease. Note: Active medical conditions that are minor or well-controlled are not exclusionary if they do not affect risk to the subject or the study results. If the effect of the condition in regard to the risk to the subject or to the study results is unclear, the Medical Monitor should be consulted.
17. Subjects with clinically relevant laboratory abnormalities at screening (eg, sodium < 130 mEq/L, alanine transaminase (ALT) or aspartate transaminase (AST) > 2.0 times the upper limit of the normal, white blood cell [WBC] count < 3,000 cells/mm3, estimated creatinine clearance < 50 mL/min, or has values for thyroid testing (free triiodothyronine (T3), free thyroxine (T4), thyroid stimulating hormone [TSH]) indicating the presence of significant thyroid dysfunction.
18. Subject has a history or presence of abnormal electrocardiogram (ECG), which in the Investigator's opinion is clinically significant or QT interval corrected for heart rate using the Fridericia method (QTcF) of ≥ 450 msec per screening ECG.
19. Subject has second or third-degree atrioventricular block that is not corrected with a pacemaker.
20. Subjects who meet the Diagnostic and Statistical Manual of Mental Disorders, 5th edition text revision defined criteria for major depressive episode within the last 6 months. Subjects with mild, chronic depression without recent hospitalization who are being maintained on a stable dose of a single antidepressant are acceptable.
21. Subject has an active suicidal plan or intent (in the Investigator's opinion) in the past 4 weeks prior to screening.
22. Subject has a history of suicide attempt in the last 2 years prior to screening.
23. Subject has other major psychiatric disorders.
24. Subjects who are not able to complete the diary in the Investigator's opinion.
25. Subject has a history of alcohol or substance abuse within 2 years prior to screening for study participation, or subjects currently using alcohol, drugs of abuse, or any prescribed or over-the-counter medication in a manner, which, in the opinion of the Investigator, indicates abuse.
26. Subject tests positive for drugs of abuse at screening. Note: Subjects with a positive drug screen for marijuana, amphetamines, opiates, or benzodiazepines, who have a documented prescription for a medical condition and are on a stable dose of this prescribed medication for at least 4 weeks prior to screening, may be eligible to participate in the study upon approval from the Medical Monitor.
27. Subject is pregnant, currently nursing, or intends to become pregnant during the study period or within 30 days of the last dose of study drug.
28. Subject has participated in any investigational study within 30 days prior to screening, as documented in subject's medical history.
29. Subject is a clinical or investigational site staff member or relative of a staff member.
30. Any other condition or circumstance that, in the opinion of the Investigator, may compromise the subject's ability to comply with the study protocol.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Director Medical Affairs, Study Chair — Sumitomo Pharma America, Inc.
Locations (55):
- United States (53):
  - University of South Alabaa Neurology Department, Mobile, Alabama
  - Banner University Medical Center Phoenix=Neuroscience Institute, Phoenix, Arizona
  - Rancho Research Institute, Inc., Downey, California
  - Neuro-Pain Medical Center, Fresno, California
  - Altman Clinical and Translational Research Institute, La Jolla, California
  - University of California-Irvine, Orange, California
  - Blue Sky Neurology, a Division of Carepoint PC, Englewood, Colorado
  - University of Connecticut School of Mwdicine -UCONN Health, Farmington, Connecticut
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Marcus Neuroscience Institute, Boca Raton, Florida
  - Infinity Clinical Research, LLC, Hollywood, Florida
  - Neurology Associates PA, Maitland, Florida
  - The Neurology Research Group, LLC, Miami, Florida
  - Laszlo J. Mate, MD, PA, North Palm Beach, Florida
  - Neurological Services of Orlando, PA, Orlando, Florida
  - Pedicatric Neurology, PA, Orlando, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - University of South Florida, Tampa, Florida
  - Vero Beach Neurology And Reasearch Institue/The MS Center of Vero Beach, Vero Beach, Florida
  - Georgia Neurology and Sleep Medicine Associates, Suwanee, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Conslutants in Epilepsy & Neurology, PLLC, Boise, Idaho
  - Northwestern Medical Group, Deparment of Neurology, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Associates in Neurology, PSC, Lexington, Kentucky
  - University of Kentucky Hospital, Chandler Medical Center, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Balijeet Shethi, MD, Waldorf, Maryland
  - Wayne State University/Detroit Medical Center, Detroit, Michigan
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Minnesota Epilepsy Group, PA, Saint Paul, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - JFK Neuroscience Institute, JFK Medical Center, Edison, New Jersey
  - Clinical Research Center of NJ (CRCNJ), Voorhees Township, New Jersey
  - NYU Winthrop Hospital, Clinical Trials Center, Mineola, New York
  - UNC Inverstigal Drug Services, Chapel Hill, North Carolina
  - The Neurological Institute, PA, Charlotte, North Carolina
  - Wake Forest Baptist Health Sciences, Department of Neurology, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Providence Medical Group-Medford Neurology, Medford, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University, Philadelphia, Pennsylvania
  - Temple University Lewis Katz School of Medicine, Philadelphia, Pennsylvania
  - Alleghany General Hospital (Allegheny Neurological Association), Pittsburgh, Pennsylvania
  - Vanderbilt Epilepsy Clinic, Nashville, Tennessee
  - Austin Epilepsy Care Center, Austin, Texas
  - Aston Ambulatory Care Center, Dallas, Texas
  - University of Texas Health Science Center at San Antonio Medical Arts and Research Center, San Antonio, Texas
  - SSM Health Dean Medical Group, Madison, Wisconsin
- Canada (2):
  - Londo Health Sciences Centre, University Hospital, London, Ontario
  - Clinique D'Épilepsie Neuro Rive-Sud, Greenfield Park, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: (arm 1) Eslicarbazepine Acetate (ESL) as first add-on to Levetiracetam or Lamotrigine)
- Arm 2: (arm 2) Eslicarbazepine Acetate (ESL) as later add-on to 1-2 Anti-epileptic drugs (AEDs)
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 44 | 58
Completed | 36 | 37
Not Completed | 8 | 21
Not completed — Adverse Event | 1 | 10
Not completed — Withdrawal by Subject | 4 | 8
Not completed — OTHER | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 44 | 58 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 38 | 53 | 91
  >=65 years | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (15.37) | 42.0 (13.83) | 42.5 (14.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 36 | 60
  Male | 20 | 22 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 37 | 51 | 88
  Unknown or Not Reported | 0 | 0 | 0
Age, Customized [Count of Participants; unit: Participants]
  > 65 years | 4 | 3 | 7
  >=18 - <=65 years | 40 | 55 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Black or African American | 8 | 16 | 24
  More than one race | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
  White | 28 | 36 | 64
  Other | 1 | 1 | 2
Country [Count of Participants; unit: Participants]
  Canada | 0 | 3 | 3
  United States | 44 | 55 | 99
Duration of Epilepsy [Count of Participants; unit: Participants]
  < 20 years | 37 | 36 | 73
  >= 20 years | 7 | 22 | 29
Number of Anti-epileptic drugs (AEDs) at Baseline [Count of Participants; unit: Participants]
  0 | 1 | 0 | 1
  1 | 42 | 21 | 63
  >=2 | 1 | 37 | 38
Use of Lamotrigine as Baseline AED [Count of Participants; unit: Participants]
  Yes | 15 | 20 | 35
  No | 29 | 38 | 67
Use of Levetiracetam as Baseline AED [Count of Participants; unit: Participants]
  Yes | 28 | 24 | 52
  No | 16 | 34 | 50
Use of Carbamazepine as Baseline AED [Count of Participants; unit: Participants]
  Yes | 0 | 5 | 5
  No | 44 | 53 | 97
Use of Valproic Acid as Baseline AED [Count of Participants; unit: Participants]
  Yes | 0 | 4 | 4
  No | 44 | 54 | 98
Use of Lacosamide as Baseline AED [Count of Participants; unit: Participants]
  Yes | 0 | 11 | 11
  No | 44 | 47 | 91
Use of Topiramate as Baseline AED [Count of Participants; unit: Participants]
  Yes | 0 | 9 | 9
  No | 44 | 49 | 93
Use of Valproate Semisodium as BL AED [Count of Participants; unit: Participants]
  Yes | 0 | 7 | 7
  No | 44 | 51 | 95
Use of Valproate All Forms as BL AED [Count of Participants; unit: Participants]
  Yes | 0 | 11 | 11
  No | 44 | 47 | 91
Rescue Medications at Baseline [Count of Participants; unit: Participants]
  Yes | 2 | 5 | 7
  No | 42 | 53 | 95
Worst Seizure Type during Baseline [Count of Participants; unit: Participants] — Population: for this outcome measure only 57 participants from arm 2 were included in the analysis
  Participants
    number analyzed (Participants) | 44 | 57 | 101
    Simple Partial | 6 | 4 | 10
    Complex Partial | 25 | 41 | 66
    Partial Evolving to Secondary Generalized | 12 | 12 | 24
    Other | 1 | 0 | 1
Baseline Height (cm) [Mean (Standard Deviation); unit: cm] | 166.9 (11.76) | 166.8 (9.73) | 166.9 (10.59)
Baseline Weight (kg) [Mean (Standard Deviation); unit: kg] | 80.23 (16.620) | 86.24 (23.841) | 83.65 (21.151)
Baseline BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 28.83 (5.694) | 30.83 (7.618) | 29.97 (6.895)
Duration of Epilepsy (years) [Mean (Standard Deviation); unit: years] | 9.4 (11.10) | 19.5 (15.90) | 15.1 (14.85)
Number of Anti-epileptic drugs (AEDs) at Baseline [Mean (Standard Deviation); unit: number of Anti-epileptic drugs (AEDs)] | 1 (0.22) | 1.7 (0.62) | 1.4 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Completing 24 Weeks Adjunctive Therapy During Maintenance Phase
Description: Phase 4 study of eslicarbazepine acetate (ESL) as adjunctive therapy in adult subjects with a diagnosis of epilepsy with Partial-onset seizures (POS). Two groups of ESL-naïve subjects will be evaluated
Time Frame: From the date of the first dose of the study drug until the completion of 24 weeks Maintenance Phase
Measure: Number; unit: participants
Groups:
- Eslicarbazepine Acetate (Arm 1): eslicarbazepine acetate (ESL) (as first add-on to Levetiracetam or Lamotrigine)
- Eslicarbazepine Acetate (Arm 2): eslicarbazepine acetate (ESL) (as later add-on to 1-2 Anti-epileptic drugs (AEDs)
Arm/Group | Eslicarbazepine Acetate (Arm 1) | Eslicarbazepine Acetate (Arm 2)
Number analyzed (Participants) | 44 | 58
participants | 36 | 37

ADVERSE EVENTS:
Time Frame: 31 weeks
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/44 | 4/58
Other Adverse Events (participants affected / at risk) | 21/44 | 36/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=44) | Arm 2 (N=58)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=44) | Arm 2 (N=58)
Diplopia (Eye disorders) | 1 (1) | 4 (7)
Nausea (Gastrointestinal disorders) | 4 (4) | 11 (13)
Vomiting (Gastrointestinal disorders) | 1 (1) | 6 (7)
Fatigue (General disorders) | 2 (2) | 9 (10)
Oedema peripheral (General disorders) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 6 (6) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Balance disorder (Nervous system disorders) | 2 (2) | 3 (3)
Coordination abnormal (Nervous system disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 8 (10) | 14 (15)
Headache (Nervous system disorders) | 5 (5) | 8 (15)
Memory impairment (Nervous system disorders) | 1 (1) | 4 (5)
Somnolence (Nervous system disorders) | 6 (6) | 6 (6)
Anxiety (Psychiatric disorders) | 1 (2) | 6 (6)
Haematoma (Vascular disorders) | 0 (0) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming withing twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish

DOCUMENTS (2):
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT03116828/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT03116828/SAP_001.pdf